CLINICAL TRIAL: NCT00858936
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of IK-1001 to Evaluate Safety, Pharmacokinetics and Proof-of-concept Efficacy for Reduction of Ischemia-Reperfusion Mediated Cardiac Injury in Subjects Undergoing Coronary Artery Bypass Graft(CABG)Surgery
Brief Title: Reduction of Ischemia-Reperfusion Mediated Cardiac Injury in Subjects Undergoing Coronary Artery Bypass Graft Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study Terminated - Company decision
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: S201
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Coronary Artery Bypass Surgery
Keywords: CABG(coronary artery bypass graft); Ischemia; Heart surgery; Heart damage
MeSH Terms: conditions — Ischemia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IK-1001 (Experimental): 6 escalating dose levels of 0.2, 0.5, 0.75, 1.0, 1.25, and 1.5 mg/kg/hr infusion for 6 hours
  Interventions: Drug: IK-1001
- Normal Saline (Placebo Comparator): 6 escalating dose levels of 0.2, 0.5, 0.75, 1.0, 1.25, and 1.5 mg/kg/hr infusion for 6 hours
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: IK-1001 — 6 escalating dose levels of 0.2, 0.5, 0.75, 1.0, 1.25, and 1.5 mg/kg/hr infusion for 6 hours
  Arms: IK-1001
Drug: Normal Saline — 6 escalating dose levels of 0.2, 0.5, 0.75, 1.0, 1.25, and 1.5 mg/kg/hr infusion for 6 hours
  Arms: Normal Saline

SUMMARY:
This clinical trial will investigate the safety and effectiveness of IK-1001 (the liquid form of sodium sulfide) when used in Coronary Artery Bypass Graft (CABG) patients to potentially reduce the damage done to the heart during surgery.

This study has 2 parts. Part 1 will first test 36 subjects at different doses (amount) of the study drug. There will be 6 different groups of 6 subjects each that will receive the study drug or a placebo. A placebo is a substance that will be prepared to look like the study drug but will contain no active ingredients. In Part 1, five subjects from each group will receive study drug (IK-1001) and one will receive a placebo. This first part of this study is also a dose (amount) escalation. This means that each group will be receiving a different dose of the study drug. The first group will receive the lowest dose, the second group will receive a slightly higher dose, and the third group a slightly higher dose until all six groups has been tested. You can not choose which group you will be in but prior to starting each new dose level, the data (information) from the previous dose level will have been reviewed by a group of qualified individuals to determine if it is safe to proceed to the next highest dose level.

Part 2 will expand the study and will treat at least 158 (and up to 632) more subjects at a dose level that has been deemed safe from information collected from Part 1. Subjects in Part 2 of the study will have a 1 in 2 (50%) chance of receiving the study drug or placebo. Whether the subject gets study drug or the placebo will be randomly assigned (like the toss of a coin).

The study drug or placebo will be given as an intravenous infusion (into the vein) for six hours while the subject is having their CABG surgery.

The subjects will be followed up for 6 months after their CABG surgery.

DETAILED DESCRIPTION:
This is a phase 2, randomized, double-blind, placebo-controlled, multicenter, dose escalation and dose-expansion, study that will evaluate safety, PK, and POC-efficacy of IK-1001 in subjects undergoing on pump CABG surgery who are at an increased risk for I/R mediated tissue damage.

Study subjects will undergo planned CABG surgery with cardiopulmonary bypass. The study will be conducted in two parts. Part 1 of the study will involve the dose escalation to evaluate safety, PK, and preliminary efficacy of IK-1001. Up to 36 eligible subjects will be enrolled into the Part 1 portion and randomized to receive either placebo (n = 6) or IK-1001 (n = 30) at 6 dose escalating levels of 0.2, 0.5, 0.75, 1.0, 1.25, and 1.5 mg/kg/hr infusion for 6 hours.

The study drug administration will begin in the operating room after the induction of anesthesia and prior to the surgical incision.

After safety, efficacy, and PK data have been evaluated in Part 1, the optimum dose will be determined and this dose will be expanded in Part 2. Initially up to 158 eligible subjects will be randomized to receive either IK-1001 or placebo at a 1:1 ratio. Part 2 aims to further establish safety, PK as well as POC efficacy.

In the event that none of the 4 primary endpoints reach at least a 15% decline as compared with placebo, the Sponsor may decide to amend the protocol to explore a higher dose. After 6 subjects have been dosed at this higher dose level, the data will be reviewed by the Sponsor or designee for safety and PK and the remaining subjects will then be enrolled. If the safety and PK data are favorable, the study will be completed at this higher dose level.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18 to 85 years of age
2. Subject is scheduled to undergo CABG surgery with cardiopulmonary bypass
3. Subjects at an increased risk for I/R mediated tissue damage: defined as subjects with ≥ 30% but ≤ 50% ejection fraction (as measured by echocardiography within 14 days of study enrollment) or who fulfill at least two of the following criteria:

   * Current or recent smoker (within last 6 months prior to screening)
   * Female
   * Diabetes mellitus (a history of diabetes, regardless of duration of disease or need for anti-diabetic agents)
   * History of non-disabling stroke, TIA, carotid endarterectomy
   * Re- CABG (H/O previous CABG surgery, on or off-pump)
   * Peripheral artery surgery or angioplasty
   * Recent MI (≥ 48 hours and ≤ 6 weeks before surgery, non STEMI and STEMI infarcts as documented in the medical records of the subject)
   * History of congestive heart failure (NYHA CHF Class III or IV)
   * Renal dysfunction: creatinine clearance ≥ 30mL/min but < 60mL/min calculated using Crockroft and Gault formula: Creatinine clearance (mL/min) = (140 - age) x weight (kg) (x 0.85 for females) (72 x serum creatinine)
   * Asymptomatic stenosis (≥ 50%) in ≥ 1 carotid artery
   * Age > 65 years

Exclusion Criteria:

1. Known sulfite allergy or sulphur drug allergy
2. Subjects who have received treatment for asthma within the past 12 months
3. Myocardial infarction occurring < 48 hours prior to surgery
4. Current cardiogenic shock, acute left ventricular rupture, ventricular septal rupture, or papillary muscle rupture
5. History of prior disabling stroke
6. Clinically relevant liver disease (defined as serum transaminases ≥ 3 x upper limit of normal for local laboratory)
7. Poorly controlled diabetes mellitus (defined as HbA1c > 9.0%)
8. Planned concomitant cardiac valve or other surgery at time of CABG
9. Planned use of thiopental during anesthesia for CABG surgery
10. All females of child bearing potential (defined as having menses without an alternative medical cause during the last 12 months). Women who are pregnant (defined as a positive serum pregnancy test), breast-feeding or lactating are also excluded.
11. Ongoing alcohol or drug abuse
12. Any underlying medical or psychiatric condition that, in the opinion of the Investigator, makes the subject an unsuitable candidate for the study
13. Subject has participated in another investigational drug or device study within 30 days prior to enrollment to the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Cardiac Troponin T | Day 1 through Day 4

SECONDARY OUTCOMES:
Mortality | Study duration
12-Lead ECG | Periodically through study duration
Urinalysis | Screening, and 6 month
Echocardiography | Screening, 3 month and 6 month
Blood Draws | Study duration
Vital Signs | Study duration
MRI | Screening, 1 month
Adverse events | Study duration
Serum levels of CK-MB | Day 1 through Day 4

CONTACTS AND LOCATIONS:
Locations (8):
- Australia (5):
  - Ashford Hospital, Ashford, South Australia
  - Flinder Medical Center, Bedford Park, South Australia
  - Austin Hospital, Heidelberg, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - St. Vincents Hospital, Melbourne, Victoria
- Canada (3):
  - Boniface General Hospital, Winnepeg, Manitoba
  - Royal Victoria Hospital - MUHC, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec